CLINICAL TRIAL: NCT07201454
Title: Holistic Evaluation of the Effects of Rehabilitative Nursing Care Practices on Frail Patients Undergoing Knee Arthroplasty and Their Caregivers
Brief Title: The Effect of Rehabilitative Nursing Care Practices on Frail Patients Undergoing Knee Arthroplasty and Their Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, İlknaz Kara, PhD Student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Ilknaz_Doktara_Tezi
Record Dates: First submitted 2025-09-11; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Knee Arthroplasty
Keywords: knee arthroplasty; fragile patient; care burden; feeling stuck; caregiver; human care theory
MeSH Terms: conditions — Caregiver Burden | interventions — Nursing Care

STUDY DESIGN:
Intervention Model Description: The study will be conducted at Erzincan Binali Yıldırım University Mengücek Gazi Training and Research Hospital between October 2025 and June 2026. The hospital has 510 beds and is planned to be conducted in 40-bed orthopedic wards I and II.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The study group will consist of patients over the age of 18 who underwent knee arthroplasty surgery at the Orthopedics and Traumatology Clinic of Erzincan Binali Yıldırım University Mengücek Gazi Training and Research Hospital, who have been hospitalized for at least four days postoperatively, and who have a score of ≥7 on the Edmonton Frailty Scale, as well as caregivers over the age of 18 who are the primary caregivers of these patients (both groups must meet criteria such as proficiency in Turkish and volunteering for the study). A total of 25 patients and 25 caregivers will participate in the experimental group.
  Interventions: Behavioral: nursing care
- Control group (No Intervention): The study group will consist of patients over the age of 18 who underwent knee arthroplasty surgery at the Orthopedics and Traumatology Clinic of Erzincan Binali Yıldırım University Mengücek Gazi Training and Research Hospital, who have been hospitalized for at least four days postoperatively, and who have a score of ≥7 on the Edmonton Frailty Scale, as well as caregivers over the age of 18 who are the primary caregivers of these patients (both groups will meet criteria such as proficiency in Turkish and volunteering for the study). A total of 25 patients and 25 caregivers will participate in the control group.

INTERVENTIONS:
Behavioral: nursing care — The first stage is the collection of quantitative data. Only quantitative data were collected from patients and caregivers in the experimental and control groups before the implementation of curative care practices based on human caring theory. The second stage includes curative care practices within the scope of the study for the experimental group. Patients and their relatives in the control group will receive routine care services provided at the clinics where the study was conducted, but no interventions will be implemented by the researchers. The third stage is the stage where patient satisfaction, caregiver burden, feelings of entrapment, and satisfaction with caregiving are assessed after the curative care practices. This stage is the final test of quantitative data and the collection of qualitative data. The fourth stage is the evaluation stage. In the final stage, data obtained from all stages will be compared, evaluated, and interpreted.
  Arms: Experimental group

SUMMARY:
This study was designed to holistically examine the effects of curative nursing care practices based on human caring theory on frail patients and their caregivers undergoing knee arthroplasty.

DETAILED DESCRIPTION:
Objective: This study was designed to thoroughly examine the effects of rehabilitative care practices based on the Human Caring Theory on the feeling of entrapment and caregiver burden of frail patients undergoing knee arthroplasty, as well as their impact on patient satisfaction.

Method: This study will be conducted as a randomized controlled experimental study with 50 frail patients and their caregivers who underwent knee arthroplasty surgery at the orthopedic ward of Erzincan Mengücek Gazi Training and Research Hospital between October 2025 and June 2026. Patients and caregivers will be assigned to experimental (25) and control (25) groups using a simple randomization method. A mixed design, randomized controlled experimental, and phenomenological study is planned to determine the effects of this study on the feeling of entrapment and caregiver burden of caregivers and on patient satisfaction.

Data collection: The Descriptive Characteristics Form will be applied to the patients' primary caregivers and their relatives. Then, the Feelings of Entrapment Scale, the Zarit Burden of Care Scale, the Caregiver Satisfaction Assessment Index (CASI-TR) and the Patient Satisfaction Assessment Form According to Watson Recovery Processes will be applied to the patients. Then, after the recovery care procedures are completed, on the 4th postoperative day, the Feelings of Entrapment Scale, the Zarit Burden of Care Scale, the Caregiver Satisfaction Assessment Index (CASI-TR) and the Patient Satisfaction Assessment Form According to Watson Recovery Processes will be applied to the patients. Then, the questions in the semi-structured interview form will be asked and their answers will be transferred as is, without any comments. They will also be audio-recorded to prevent data loss and to ensure that the responses can be listened to again by the researcher later. The Feelings of Entrapment Scale, the Zarit Caregiver Burden Scale, and the Caregiver Satisfaction Assessment Index (CASI-TR) will be administered to the primary caregivers and patients in the control group on Day 4. The Patient Satisfaction Assessment Form will be administered to the patients based on Watson Improvement Processes.

Original Value: No studies have been found in the literature that evaluate the theoretical basis of caregiver care for frail patients undergoing knee arthroplasty surgery, their satisfaction with caregiving, the impact of feeling entrapment, or patient satisfaction. In this respect, the project has unique value and will contribute scientifically to national and international literature. If successful, it is expected to introduce holistic nursing care practices to the field regarding the care of frail patients undergoing knee arthroplasty surgery, which presents significant challenges for caregivers. In this respect, the project has unique value.

Expected Outcome: If the project is successful, it will reduce anxiety and caregiver burden in patients' relatives and increase patient-family interaction, contributing to improved patient care and economic efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Speak and understand Turkish
* Be over 18 years of age
* Have a patient they care for undergoing knee arthroplasty
* Be a caregiver for a frail patient who scores 7 or higher on the Edmonton Frailty Scale
* Provide primary care for the patient
* Voluntarily participate in the study

Exclusion Criteria:

Patient-related exclusion criteria:

* Developing serious surgical complications (e.g., infection, embolism, prosthesis rejection, etc.) after knee arthroplasty
* Admission to the intensive care unit after surgery
* Re-surgery during the postoperative period
* Death of the patient during the study
* Voluntary withdrawal from the study or lack of communication

Caregiver-related exclusion criteria:

* Transfer of caregiving role to another person after the study begins
* Caregivers experiencing a physical or psychological health problem that would prevent them from continuing the study
* Caregivers refusing to continue the study or lack of communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The effect of healing care on caregiver entrapment will be measured with the Feeling of Entrapment Scale, preoperatively and on the 4th postoperative day. Outcome is the change in total score. | 4 days before and 4 days after application
The effect of therapeutic care on caregiver burden will be measured with the Zarit Caregiver Burden Scale (0-88), preoperatively and on the 4th postoperative day. Outcome is the change in total score. | 4 days before and 4 days after application
The effect of healing care on caregiver satisfaction will be measured with the Caregiver Satisfaction Index (1-5), preoperatively and on the 4th postoperative day. Outcome is the change in satisfaction score. | 4 days before and 4 days after application
The effect of therapeutic care on patient satisfaction will be measured with the Patient Satisfaction Form based on Watson's Healing Processes (0-100), preoperatively and on the 4th postoperative day. Outcome is score change. | 4 days before and 4 days after application

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk, Zubeyde Hanim St. No: 10, 24180 Erzincan Center/Erzincan, Erzincan, Erzincan 24180, Erzincan, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No